CLINICAL TRIAL: NCT06635486
Title: Adaptation of an Open Source Cognitive Behavioral Treatment Protocol Designed to Improve Mental Health in Forcibly Displaced Populations
Brief Title: Improving Mental Health in Forcibly Displaced Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-45280; 1K23MH127308 (NIH)
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Post Traumatic Stress Disorder; Depression
Keywords: Venezuelan migrants; Cognitive behavioral intervention (CBT); Culturally adapted; Lay providers; Feasibility; Acceptability
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Depression | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the intervention (n = 60) or wait list control (n = 30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants randomized to this arm will receive the CBT adapted intervention.
  Interventions: Behavioral: Adapted cognitive-behavioral (CBT) intervention
- Wait list control arm (No Intervention): Participants randomized to this arm will be placed on a wait list for the CBT adapted intervention.

INTERVENTIONS:
Behavioral: Adapted cognitive-behavioral (CBT) intervention — The intervention is 6-12 sessions, depending on the symptom presentation of the participant. The weekly sessions last 60 minutes and will be delivered remotely and individually via Meet or a similar platform by trained lay providers. Intervention methods include cognitive re-structuring, behavioral activation, exposure to memories and situations, problem solving, and emotional regulation.
  Other Names: A culturally adapted transdiagnostic CBT intervention
  Arms: Intervention arm

SUMMARY:
This project aims to improve mental health support for Venezuelan migrants living in Lima, Peru, who often face challenges like anxiety, depression, and post-traumatic stress disorder (PTSD). Since 2015, millions of Venezuelans have fled their country due to a severe humanitarian crisis, including extreme inflation, food shortages, and political unrest. Many of these individuals now live in Peru, where they struggle to access mental health services.

A new type of intervention that is both evidence-based and culturally adapted to meet the specific needs of Venezuelan migrants is the focus of this research. The intervention is designed to be delivered by trained lay providers-people from the community who have received special training but are not professional mental health workers. The intervention consists of 6 to 12 weekly online sessions, each lasting about an hour. These sessions will cover various therapeutic techniques, including cognitive restructuring (changing negative thought patterns), behavioral activation (encouraging positive activities), and emotional regulation (managing feelings). The sessions will be conducted remotely, allowing participants to join from the comfort of their homes.This approach is intended to make mental health care more accessible and relatable for migrants, who may feel more comfortable receiving help from someone who understands their cultural background and experiences.

DETAILED DESCRIPTION:
To assess the effectiveness of this intervention, 90 participants will be assigned into two groups: one that receives the intervention and another that will be on a waitlist for later participation. The investigators will measure changes in mental health symptoms using validated questionnaires throughout the study and at follow-up intervals. Participants will also provide feedback on their experience, providing information on how acceptable and feasible this approach is.

The three goals of the trial are:

1. Efficacy: To determine if the intervention effectively reduces symptoms of anxiety, depression, and PTSD among participants.
2. Feasibility and Acceptability: To evaluate how practical and well-received the intervention is by both participants and providers.
3. Understanding Moderating Factors: To explore how individual experiences related to migration and integration affect the success of the intervention.

By focusing on a vulnerable population that often lacks access to traditional mental health resources, this project aims to provide valuable insights into effective mental health strategies for forcibly displaced individuals. If successful, the findings could help inform community leaders, non-governmental organizations (NGOs), and health care providers about how to better support Venezuelan migrants and potentially other migrant groups facing similar challenges in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* have Venezuelan nationality
* have arrived in Lima in years 2014 to the present
* be 18 years of age or older

In addition, in order to be eligible to participate in this study, an individual must meet one of the following criteria:

* score 10 points or more at the Patient Health Questionnaire (PHQ-9) or
* score 10 points or more at the General Anxiety Disorder (GAD-7) or
* have a history of trauma exposure as listed in the Life Events Checklist (LEC-5) and score 31 points or more in the PTSD Checklist (PCL-5)

Exclusion Criteria:

An individual is excluded from the study if they respond positively to one or more of the following questions during screening:

* Suicidal ideation: "When someone feels as upset as you do, they may have thoughts that life isn't worth living. What thoughts have you had like this?"
* Homicidal ideation: "When someone feels as upset as you do, they may have thoughts about hurting the person who has upset or hurt them. What thoughts have you had like this?"
* Psychosis: "Do you have a diagnosis of psychosis or schizophrenia?"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Throughout the study (on average 10 months for each participant). Outcome will be assessed every 2 weeks during the intervention (on average 3 months long), and after completion of the intervention at 1 month, 3 months, and 6 months follow-up
  Anxiety will be assessed using the 7-item Generalized Anxiety Disorder (GAD-7). Each item is scored from 0 to 3, where 0= Not at all and 3= Nearly every day, with a range of scores from 0 to 21. The interpretation of scores are: 0 - 4: Minimal anxiety, 5 - 9: Mild anxiety, 10 -14: Moderate anxiety, and 15+: Severe anxiety.
Depression | Throughout the study (on average 10 months for each participant). Outcome will be assessed every 2 weeks during the intervention (on average 3 months long), and after completion of the intervention at 1 month, 3 months, and 6 months follow-up
  Depression will be assessed using the 9-item Patient Health Questionnaire (PHQ-9). Each item is scored from 0 to 3, where 0= Not at all and 3= Nearly every day, with a range of scores from 0 to 27. The interpretation of scores are: 0-4: No or minimal depression, 5-9: Mild depression, 10-14: Moderate depression, 15-19: Moderately severe depression, 20-27: Severe depression.
Post Traumatic Stress Disorder (PTSD) | Throughout the study (on average 10 months for each participant). Outcome will be assessed every 1 week during the intervention (on average 3 months long), and after completion of the intervention at 1 month, 3 months, and 6 months follow-up
  PTSD will be assessed with the PTSD Checklist (PCL-5). Participants will rate how bothered they have been in the past month for 20 items where each is scored from 0 to 4, where 0=Not at all to 4=Extremely. The range of scores is 0 to 80, and higher scores are associated with higher PTSD symptoms.
Traumatic Life Events | Throughout the study (on average 10 months for each participant). Outcome will be assessed every 2 weeks during the intervention (on average 3 months long), and after completion of the intervention at 1 month, 3 months, and 6 months follow-up
  The Life Events Checklist for DSM-5 (LEC-5) will be used to assess traumatic life events. It does not have a formal scoring protocol or interpretation, other than to identify if a person has experienced any of the listed events. The LEC-5 does not provide a total or composite score.

SECONDARY OUTCOMES:
Recruitment feasibility | Throughout the study (on average 10 months for each participant). Outcome will be assessed for each participant one time at the start of the study.
  Recruitment feasibility is defined as the percent of eligible participants who enroll in the study.
Retention | Throughout the study (on average 10 months for each participant). Outcome will be assessed every 1 week during the intervention (on average 3 months long), and after completion of the intervention at 1 month, 3 months, and 6 months follow-up
  Retention is defined as the number of participants who completed all study visits and follow-up assessments.
Fidelity | Throughout the intervention (on average 3 months for each participant). Outcome will be assessed every 1 week during the intervention.
  Fidelity is defined by the adherence and competence scores (0 to 10) from research staff assessment of audio recorded sessions. Higher scores are associated with greater fidelity.
Provider perception of participant satisfaction | Throughout the intervention (on average 3 months for each participant). Outcome will be assessed every 1 week during the intervention.
  Defined as the satisfaction of the participant in the session's helpfulness, enjoyment and relevance (0 to 10), with higher scores being associated with greater satisfaction.
Provider perception of participants' future use | Throughout the intervention (on average 3 months for each participant). Outcome will be assessed every 1 week during the intervention.
  Defined as participants' plans to use material learned in the future (Yes/No)
Participant perception of participant satisfaction | Throughout the intervention (on average 3 months for each participant). Outcome will be assessed every 1 week during the intervention.
  Defined as direct participant report of their satisfaction of the session's helpfulness, enjoyment and relevance (0 to 10), with higher scores being associated with greater satisfaction.
Participant perception of future use | Throughout the intervention (on average 3 months for each participant). Outcome will be assessed every 1 week during the intervention.
  Defined as participants' plans to use material learned in the future (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Haley Carroll, PhD MS, Principal Investigator — Boston Medical Center, BUCA School of Medicine
Locations (1):
- Universidad del Pacifico, Lima, Peru

IPD SHARING:
Plan to Share IPD: No